CLINICAL TRIAL: NCT02621372
Title: Correlation of Platelets Count With Endoscopic Findings in a Cohort of Egyptian Patients With Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Hepatology and gastroenterology dept., tanta university, M.D., Principle investigator, Tanta University
Organization: Tanta University (Other)
Other Study IDs: non invasive diagnosis of EV
Record Dates: First submitted 2015-11-27; First posted 2015-12-03 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Platelet Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: platelet count — Correlation of esophageal varices with platelet count

SUMMARY:
Portal hypertension is a common complication of liver cirrhosis that can lead to development of esophageal varices (EV). They are abnormally dilated veins within the wall of the esophagus that lead to haemorrhage (1). Majority of patients with cirrhosis will develop EV at some point, and about third of these patients will have at least one bleeding episode because of rupture of a varix . For this reason, screening endoscopy for detection of the presence of EV should be part of the diagnostic work-up in patients with cirrhosis. This is a very important preventive step for identification of those patients with variceal bleeding risk and furthermore, identification of patients in urgent need for prophylactic treatment.

All guidelines stress on screening endoscopy for early detection of EV in cirrhotic patients with portal hypertension. However this approach is limited by its invasiveness and cost effectiveness issues of screening endoscopy .

DETAILED DESCRIPTION:
Recent research has focused on the use of noninvasive methods to detect patients with the intention of avoiding endoscopy in low-risk cases . Thrombocytopenia (platelet count < 150,000/μl) is a common complication in patients of chronic liver disease (CLD) . So, the investigators in this research formulated this study to determine whether platelet count can predict the presence of EV or varices which need prophylactic therapy (medium or large size EV) in a cohort of Egyptian patients with liver cirrhosis and can identify patients with the intention of avoiding endoscopy in low-risk cases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis based on history, physical examination, laboratory tests, ultrasound scans and liver biopsy in some occasion.

Exclusion Criteria:

* Hepatocellular carcinoma.
* Portal vein thrombosis.
* Parenteral drug addiction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 110 cirrhotic patients were included
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with esophageal varices and have low platelet count | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-Elsalam, Principal Investigator — Tanta university hospital
Locations (1):
- Tropical medicine dept.-Tanta university hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided